CLINICAL TRIAL: NCT05925738
Title: Positron Emission Tomography/ Computed Tomography (PET/CT) Based Deep Learning Signature for Predicting Aggressive Histological Pattern in Resected Non-small Cell Lung Cancer
Brief Title: Deep Learning Signature for Predicting Aggressive Histological Pattern in Resected Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Ningbo No.2 Hospital (Other); Zunyi Medical College (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Chang Chen, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: DLAHP
Record Dates: First submitted 2023-05-12; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Non-small Cell Lung Cancer; Spread Through Air Space; Visceral Pleural Invasion; Lymphovascular Invasion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET/CT-based Deep Learning Signature — Deep Learning Signature Based on PET-CT for Predicting the Aggressive Histological Pattern in Resected Non-small Cell Lung Cancer

SUMMARY:
The purpose of this study is to evaluate the performance of a PET/ CT-based deep learning signature for predicting aggressive histological pattern in resected non-small cell lung cancer based on a multicenter prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

(1) Participants scheduled for surgery for radiological finding of pulmonary lesions from the preoperative thin-section CT scans; (2) Pathological confirmation of primary NSCLC; (3) Age ranging from 20-75 years; (4) Obtained written informed consent.

Exclusion Criteria:

(1) Multiple lung lesions; (2) Poor quality of PET-CT images; (3) Participants with incomplete clinical information; (4) Participants who have received neoadjuvant therapy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Resected Stage I-III Non-small Cell Lung Cancer
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve | 2023.5.1-2023.10.31
  The area under the receiver operating characteristic curve (ROC) of the deep learning model in predicting the presence or absence of the aggressive histological pattern. The aggressive histological pattern includes spread through air space (STAS), visceral pleural invasion (VPI), and lymphovascular invasion (LVI). And the model will output all predictive values (presence or absence) of the three kinds of aggressive histological patterns.

SECONDARY OUTCOMES:
Sensitivity | 2023.5.1-2023.10.31
  The sensitivity of the deep learning model in predicting the presence or absence of the aggressive histological pattern. The aggressive histological pattern includes spread through air space (STAS), visceral pleural invasion (VPI), and lymphovascular invasion (LVI). And the model will output all predictive values (presence or absence) of the three kinds of aggressive histological patterns.

OTHER OUTCOMES:
Specificity | 2023.5.1-2023.10.31
  The specificity of the deep learning model in predicting the presence or absence of the aggressive histological pattern. The aggressive histological pattern includes spread through air space (STAS), visceral pleural invasion (VPI), and lymphovascular invasion (LVI). And the model will output all predictive values (presence or absence) of the three kinds of aggressive histological patterns.
Positive predictive value | 2023.5.1-2023.10.31
  The positive predictive value of the deep learning model in predicting the presence or absence of the aggressive histological pattern. The aggressive histological pattern includes spread through air space (STAS), visceral pleural invasion (VPI), and lymphovascular invasion (LVI). And the model will output all predictive values (presence or absence) of the three kinds of aggressive histological patterns.
Negative predictive value | 2023.5.1-2023.10.31
  The negative predictive value of the deep learning model in predicting the presence or absence of the aggressive histological pattern. The aggressive histological pattern includes spread through air space (STAS), visceral pleural invasion (VPI), and lymphovascular invasion (LVI). And the model will output all predictive values (presence or absence) of the three kinds of aggressive histological patterns.
Accuracy | 2023.5.1-2023.10.31
  The accuracy of the deep learning model in predicting the presence or absence of the aggressive histological pattern. The aggressive histological pattern includes spread through air space (STAS), visceral pleural invasion (VPI), and lymphovascular invasion (LVI). And the model will output all predictive values (presence or absence) of the three kinds of aggressive histological patterns.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Ningbo HwaMei Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No